CLINICAL TRIAL: NCT04150393
Title: Safety Phase I Evaluation of MaaT033, a Lyophilized Full-ecosystem Gut Microbiota Delayed-release Capsule, In HeMatOlogy Malignant Patients Under iNtensive Chemotherapy (CIMON)
Brief Title: Safety and Tolerability Evaluation of MaaT033
Acronym: CIMON
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MaaT Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: MPOH05
Record Dates: First submitted 2019-10-25; First posted 2019-11-04 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Hematologic Diseases; Chemotherapy Effect
Keywords: microbiota; microbiotherapy
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Intervention Model Description: 3+3 design dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MaaT033 treatment (Experimental): A Lyophilized Full-ecosystem Gut Microbiota Delayed-release Capsule
  Interventions: Drug: MaaT033 capsule

INTERVENTIONS:
Drug: MaaT033 capsule — Oral capsule

SUMMARY:
Richness and diversity of gut microbiota are increasingly found to be associated with cancer outcomes. Moreover, an adequately responsive immune system seems to rely on the existence of a functioning gut ecosystem that includes the microbiota and its natural environment.

Cancer by itself, but also cancer treatments - in particular chemotherapy - induce gut dysbiosis, impair the constant reparation mechanisms of the gut epithelium, disrupt immune homeostasis, and stunt immune responsiveness.

The objective of MaaT033 is to (1) prevent the decay of the gut ecosystem (dysbiosis) to preserve immune homeostasis, (2) restore and optimize the gut ecosystem to full functionality including its role in repairing the gut epithelium and healthy gut barrier, and (3) maintain a restored gut ecosystem and fully functional immune homeostasis.

Restoring the full gut ecosystem and its associated microbiota could become an important therapeutic option to improve clinical outcomes and control adverse events of conventional approaches, including immunotherapy in cancer patients.

As a first step, MaaT033 capsules containing lyophilized, pooled, full-ecosystem microbiota in its natural environment are to be tested for their safety and tolerability in hematological malignant patients, who are exposed to intensive rounds of chemotherapy and antibiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Age ≥ 18 years
3. Patients diagnosed with AML defined according to WHO 2016 criteria with ≥20% leukemic blasts in the bone marrow or with high- risk myelodysplastic syndrome, receiving intensive chemotherapy
4. Patients healthy enough to likely receive their consolidation or second cycle of chemotherapy after induction chemotherapy
5. Patients healthy enough to likely receive HSCT
6. Informed written consent
7. Patient recovered from neutropenia

Exclusion Criteria:

1. Acute promyelocytic leukemia (AML-M3)
2. AML secondary to myeloproliferative disorder or chronic myelomonocytic leukemia (CMML)
3. Acute myeloid leukemia BCR-ABL1+
4. Active CNS leukemia
5. Patients with a life expectancy of <70 days according to investigator's opinion, or subject to therapeutic limitations
6. Confirmed or suspected intestinal ischemia
7. Confirmed or suspected toxic megacolon or gastrointestinal perforation
8. Active uncontrolled infection according to the attending physician
9. Any gastro-intestinal bleeding in the past 3 months
10. Any history of gastro-intestinal surgery in the past 3 months
11. Any history of inflammatory bowel disease
12. Any counter-indication to swallow capsules
13. Enrollment in another trial that may interfere with this study
14. Known allergy or intolerance to trehalose, maltodextrin or PEG
15. Women of childbearing potential without efficient contraceptive protection
16. Pregnant or breastfeeding
17. Patients with EBV-negative serology
18. Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
19. Exclusion period of a previous study
20. Administrative or legal supervision
21. Confirmed positive result to SARS-CoV-2 nasopharyngeal test at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Occurrence of MaaT033-related, treatment-emergent (serious) adverse events, grade >3, as assessed by CTCAE v4.0 | From treatment start (V1, end of aplasia) to the end of the study (end of consolidation or up to 10 weeks)
  Evaluation of safety and tolerability of MaaT033 in patients with hematologic malignancies

SECONDARY OUTCOMES:
Dose regimen evaluation | From treatment start (V1, end of aplasia) to the end of the study (end of consolidation or up to 10 weeks)
  Activity assessment of the different dose regimens defined as bacterial "engraftment" of the product

CONTACTS AND LOCATIONS:
Overall Officials: Christian Recher, Pr, Principal Investigator — IUCT
Locations (4):
- France (4):
  - CHU Angers, Angers
  - CHU Nice, Nice
  - APHP St Antoine, Paris
  - IUCT, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malard F, Thepot S, Cluzeau T, Carre M, Lebon D, Bories P, Legrand O, Schwarz M, Loschi M, Meunier M, Joris M, Gasc C, Jouve J, Levast B, Plantamura E, Prestat E, Sabourin A, Gaugler B, Dore J, Recher C, Mohty M. Gut microbiota restoration with oral pooled fecal microbiotherapy after intensive chemotherapy: the phase 1b CIMON trial. Blood Adv. 2025 Aug 12;9(15):3739-3749. doi: 10.1182/bloodadvances.2024015571. PMID 40197991